CLINICAL TRIAL: NCT05077748
Title: An 18-year Follow-up Study on Obstructive Sleep Apnoea in a Population-based Cohort
Brief Title: An 18-year Follow-up Study on OSA in a Population-based Cohort
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Clinical Professional Consultant, Department of Paediatrics, Chinese University of Hong Kong
Other Study IDs: FUOSA 3.1
Record Dates: First submitted 2021-10-02; First posted 2021-10-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Epidemiology; Natural History; Obstructive Sleep Apnea; Cardiovascular Complication; Neurocognitive Dysfunction
Keywords: Obstructive sleep apnea; Sleep disordered breathing; Hypertension; Cardiovascular complication; Neurocognitive dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognition Disorders; Sleep Apnea Syndromes; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fasting blood samples will be taken from participants with venipuncture. The sample will be sent for biochemical measurements including lipid profile (Total cholesterol, total glycerides, high-density lipoprotein-cholesterol, low-density lipoprotein cholesterol) and serum glucose in the University Pathology Service. Plasma will also be collected in EDTA anticoagulant tubes, pre-processed and frozen at -80 degree Celsius for future analysis. Because of budget limitation, further blood test analysis is not included in the current proposal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Our research team has established a polysomnography (PSG) quantified population-based paediatric sleep cohort in 2003 for a childhood OSA prevalence study. Subjects were recruited from 13 randomly selected primary schools. All subjects from this original cohort will be invited to join this 18-year follow-up study to repeat the following data collection: questionnaires, anthropometric measurement, sleep study, 24-hour ambulatory blood pressure (ABP) measurement, echocardiography and neurocognitive assessment.

DETAILED DESCRIPTION:
Our research team has established a polysomnography (PSG) quantified population-based paediatric sleep cohort in 2003 for a childhood OSA prevalence study. Subjects were recruited from 13 randomly selected primary schools. In each school, two randomly chosen classes from each grade were invited to participate. In the first phase, all parents of children in the randomly selected schools were invited to attend an education forum during which full explanation of the purpose and flow of the study was given. An envelope containing a validated parent proxy OSAS screening questionnaire and consent was then distributed to parents within a week after the forum. From our previous research, a composite symptom score (summation of the scores of these three questions) of 7 or more has 75.4% sensitivity and 80.5% specificity, compared with polysomnography, to detect OSAS among children aged 5-15 years who had attended our paediatric clinics. Children with a composite symptom score of less than 7 were assigned a computer-generated random number and were invited as a control group with a ratio of 1:2 in the second phase. All children belonging to the high risk of OSAS group and the randomly selected subjects at low risk of OSAS were invited to participate the baseline epidemiological study. In total 619 children aged 5-13 years underwent detailed assessments including anthropometric measurements, airway examination, ambulatory blood pressure recording and overnight PSG. 67 children had moderate-to-severe OSA (obstructive apnoea hypopnoea index, OAHI ≥5/h), 199 had mild OSA (OAHI 1 to <5/h), 103 were primary snorers (OAHI <1/h but snore ≥3 nights per week in the past 12 months) and 250 were normal controls (OAHI <1/h and snore <3 nights per week in the past 12 months).(1) All subjects from this original cohort will be invited to join this 18-year follow-up study to repeat the following data collection: questionnaires, anthropometric measurement, sleep study, 24-hour ambulatory blood pressure (ABP) measurement, echocardiography and neurocognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

- Subjects participants from the 2003 cohort

Exclusion Criteria:

* Neuromuscular disease
* Pathological central apnoea
* Severe chronic lung disease with documented hypoxaemia or awake oxygen saturation <92%
* Chronic respiratory failure (unrelated to OSA)
* Acquired upper airway disease/obstruction
* Craniofacial abnormalities (e.g. secondary to trauma and malignancy)

Other arrangement:

* Subjects who have any respiratory illness within 2 weeks of the scheduled follow-up visit will have their assessment re-arranged until they have fully recovered.
* Subjects taking medications that may affect sleep, upper airway patency or blood pressure (for example sedatives, stimulants, antihistamines, and cough medicine) within a week from recruitment will also be rescheduled to participate when they are free from medication use for at least 2 weeks.
* Subjects with hypertension and are on anti-hypertensive therapy are allowed to continue on their medication and the information will be obtained and recorded during data collection.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In our current proposal, subjects from the 2003 cohort will be invited to join this follow-up study. Written consent will be obtained from the participants. The study protocol will be conducted in compliance with the Declaration of Helsinki. Ethics approval will be obtained from the Clinical Research Ethics Committee of the Joint Chinese University of Hong Kong - New Territories East Cluster.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
OSA status at 18-year follow-up visit | Through study completion, an average of 2 years
  OSA status of the participants at the 18-year follow-up visit

SECONDARY OUTCOMES:
Factors associated with the persistence or the development of OSA in adulthood | Through study completion, an average of 2 years
  Factors associated with the persistence or the development of OSA in adulthood
Ambulatory blood pressure parameters at 18-year follow-up visit | Through study completion, an average of 2 years
  Ambulatory blood pressure parameters as measures of long-term cardiovascular participants of children who had OSA compared to those without OSA
Echocardiographic parameters at 18-year follow-up visit | Through study completion, an average of 2 years
  Echocardiographic parameters as measures of long-term cardiovascular outcomes of participants who had OSA compared to those without OSA
Neurocognitive function at 18-year follow-up visit | Through study completion, an average of 2 years
  Neurocognitive function outcomes as measures of long-term neurocognitive outcomes of participants who had OSA compared to those without OSA

CONTACTS AND LOCATIONS:
Overall Officials: Ching Ching, Kate Dr. CHAN, Study Director — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available at this moment.